CLINICAL TRIAL: NCT06008301
Title: Comparing Impact of Contrast-enhanced Mammography (CEM) to Breast MRI on Barriers to Breast Cancer Treatment
Brief Title: Comparing Breast Magnetic Resonance Imaging (MRI) and Contrast-enhanced Mammography (CEM)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study never started as the PI left the insitution before IRB approval.
Sponsor: Boston Medical Center (Other)
Collaborators: Breast Cancer Alliance (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-44009
Record Dates: First submitted 2023-08-18; First posted 2023-08-23 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer Female
Keywords: Contrast enhanced mammography (CEM); Breast MRI; Financial costs; Time costs; State-trait anxiety inventory (STAI)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Consent for the entire study (Experimental): Participants with a newly diagnosed breast cancer and recommended for enhanced imaging will be randomly assigned to either CEM or MRI and take the State-Trait Anxiety Inventory (STAI) before and after imaging.
  Interventions: Other: State-Trait Anxiety Inventory (STAI)
- Consent only for the STAI (Active Comparator): Participants with a newly diagnosed breast cancer and recommended for enhanced imaging but who cannot or choose not to be randomly assigned to CEM or MRI but they consent to take the State-Trait Anxiety Inventory (STAI) before and after imaging.
  Interventions: Other: State-Trait Anxiety Inventory (STAI)

INTERVENTIONS:
Other: State-Trait Anxiety Inventory (STAI) — The State-Trait Anxiety Inventory (STAI) has 20 items for assessing trait anxiety and 20 for state anxiety.

SUMMARY:
The investigators will study the financial, time, and psychologic benefit of Contrast Enhanced Mammography (CEM) compared with Magnetic Resonance Imaging (MRI) for breast cancer evaluation and ultimately encourage practices and referring providers to use it more routinely in practice.

Specific research objectives are to:

* determine financial costs of performing a CEM to breast MRI
* compare time costs involved with CEM to breast MRI
* compare psychologic costs involved with CEM to breast MRI.

ELIGIBILITY:
Inclusion Criteria:

* Age > or equal to 30 years
* Clinically eligible for CEM or breast MRI
* Newly diagnosed cancer

Exclusion Criteria:

* Pregnant as verified by patient report. Given that this test is being performed for clinical purposes, the determination of pregnancy status will be resolved via the standard clinical pathway.

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-04 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Institutional financial costs | 24 months
  True institutional costs will be calculated using time-driven activity based costing (TDABC) methodology to estimate the capacity cost rate (CCR, defined as cost per unit time in dollars per minute for personnel, equipment, and fixed equipment) and total cost (TC, defined as the sum of CCR per resource multiplied by time utilization and added to cost of consumable materials) for MRI and CEM.
Patient financial costs | 24 months
  Patient costs will be determined by capturing insurance coverage and hospital-provided patient charges.
Time from diagnosis to imaging modality (CEM or MRI) | 24 months
  Time will be measured in days and abstracted from medical records.
Time from diagnosis to first treatment | 24 months
  Time will be measured in days and abstracted from medical records.
Number of patient visits generated from the imaging modality | 24 months
  Number of patient visits generated from the imaging modality will be abstracted from medical records.
Psychologic costs to patients | 24 months
  The State-Trait Anxiety Inventory (STAI) has 20 items for assessing trait anxiety and 20 for state anxiety. All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). Higher scores indicate greater anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Jordana Phillips, MD FSBI, Principal Investigator — Boston Medical Center, Dept of Radiology

IPD SHARING:
Plan to Share IPD: No